CLINICAL TRIAL: NCT06647875
Title: The Impact of Complementary Feeding Education Given to Fathers on Father-Infant Relationship and Infant Feeding Behavior
Brief Title: Complementary Feeding Education & Fathers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Oyku Ozboru Askan, Assistant Professor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IUICH_01
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Nutrition, Healthy; Father-Child Relations
Keywords: complementary feeding, father-child relationship

STUDY DESIGN:
Intervention Model Description: After being informed about the study and giving written consent, the parents of the infants included in the study were stratified according to the father's education level, birth order of the child, and self-efficacy scale scores, and then in order of admission to hospital assigned to the study and control groups.
Who Masked: Participant
Masking Description: participants do not know which group they are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): During their infants' 6-month check-up, parents will be administered a demographic survey, the Karitane Parental Self-Efficacy Scale, the Behavioral Pediatric Feeding Assessment Scale, the Edinburgh Postnatal Depression Scale, and the Generalized Anxiety Disorder-7 scale. The Father-Infant Bonding Scale will be administered exclusively to fathers during the same visit. Subsequently, both mothers and fathers in this group will receive complementary feeding education.
  Interventions: Behavioral: Complementary Feeding Education
- Control Group (Active Comparator): During their infants' 6-month check-up, parents will be administered a demographic survey, the Karitane Parental Self-Efficacy Scale, the Behavioral Pediatric Feeding Assessment Scale, the Edinburgh Postnatal Depression Scale, and the Generalized Anxiety Disorder-7 scale. The Father-Infant Bonding Scale will be administered exclusively to fathers during the same visit. Subsequently, only mothers in this group will receive complementary feeding education.
  Interventions: Behavioral: Complementary Feeding Education

INTERVENTIONS:
Behavioral: Complementary Feeding Education — This training program has been designed in accordance withWHO Guideline for Complementary Feeding of Infants and Young Children 6-23 Months of Age. The training will be delivered both in-person and via tablet, and will be supported by infographics and visuals created using WHO Guideline for Complementary Feeding of Infants and Young Children 6-23 Months of Age and the "Basic Information for Families on Child Health and Safety in the First 5 Years" booklet published by the Child Health Association, specifically the section on "Healthy Eating." At the end of the training, participants will be provided with a booklet containing the "Healthy Eating" section of the Child Health Association's booklet.

SUMMARY:
The aim of this study is to investigate the effect of complementary feeding education provided to fathers on father-infant bonding and infant feeding behavior. To assess father-infant bonding, the study will use the Father-Infant Bonding Scale and the Karitane Parenting Self-Efficacy Scale. For assessing infant feeding behavior, the Behavioral Pediatric Feeding Assessment Scale will be employed. These scales will be administered to participants both before and 3 months after the training.

DETAILED DESCRIPTION:
The study aims to investigate the effects of complementary feeding education provided to fathers on father-infant bonding and infant feeding behavior.

This prospective, non-randomized controlled study was conducted with the parents of 6-month-old infants followed up at the Child Health Monitoring Polyclinic of the Department of Social Pediatrics, Department of Child Health and Diseases, Istanbul Faculty of Medicine, Istanbul University. After being informed about the study and giving written consent, the parents of the infants included in the study were stratified according to the father's education level, birth order of the child, and self-efficacy scale scores, and then in order of admission to hospital assigned to the study and control groups. Infants born at term, exclusively breastfed for the first 6 months, without chronic diseases, and whose parents lived together were included in the study. Exclusion criteria included: food allergy, developmental milestones not appropriate for age, known swallowing dysfunction, psychiatric illness of either parent, a chronic illness in a sibling, adoption, and refusal to give consent.

During the 6-month check-up, parents who agreed to participate in the study completed a demographic questionnaire, the Karitane Parenting Self-Efficacy Scale (KPSCS), the Behavioral Pediatric Feeding Assessment Scale (BPFAS), the Edinburgh Postnatal Depression Scale (EPDS), and the Generalized Anxiety Disorder-7 (GAD-7) scale. The Father-Infant Bonding Scale (FIB Scale) was administered only to fathers during the same examination.

In the study group, both mothers and fathers received complementary feeding education, while in the control group, only mothers received the education. The education was based on the WHO Guideline for Complementary Feeding of Infants and Young Children 6-23 Months of Age and was delivered both in-person and via tablet. To make the education more understandable, infographics and visuals prepared using the WHO Guideline for Complementary Feeding of Infants and Young Children 6-23 Months of Age and the Basic Information for Families on Child Health and Safety in the First 5 Years booklet of the Child Health Association. At the end of the training, participants were given a booklet containing the infographics from the "Basic Information for Families on Child Health and Safety in the First 5 Years" booklet of the TChild Health Association.

At the 9-month follow-up, the KPSCS, EPDS, BPFAS, and GAD-7 scales were administered to both mothers and fathers, and the FIB Scale was administered only to fathers.

ELIGIBILITY:
Inclusion Criteria:

* Infant born at term (>37 weeks)
* Exclusively breastfed for the first 6 months and has completed postnatal month 6
* Both parents live together
* Infant feeding is done by mother, mother and father together, grandmother, or caregiver
* Infant has no chronic disease

Exclusion Criteria:

* Infant has a chronic disease
* Infant has a known food allergy
* Developmental milestones are not age-appropriate
* Known swallowing dysfunction
* Either parent has a psychiatric illness
* Sibling has a chronic disease if applicable
* Child is adopted
* Consent is not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Karitane Parenting Self Confidence Scale | 6-month and 9-month infant check-ups
  The Karitane Parenting Self-Confidence Scale (KPSCS), developed by Crncec et al. in 2008 and adapted into Turkish by Yılmaz and Oskay in 2021, is a 15-item scale designed to assess parenting self-efficacy in parents of infants aged 0-12 months. Each item is rated on a 4-point Likert scale ranging from 0 (No, not at all) to 3 (Yes, very often). Higher total scores indicate greater parenting self-efficacy.
Paternal-infant attachment scale | 6-month and 9-month infant check-ups
  The Father-Infant Bonding Scale (FIB Scale), developed by Condon et al. in 2008 and adapted into Turkish by Güleç et al. in 2010, is a 19-item scale designed to measure the strength of the father-infant bond. The scale consists of three subscales: patience and tolerance, enjoyment of interaction, and love and pride. Each item is rated on a 5-point Likert scale. The scale includes reverse-scored items (items 4, 5, 7, 8, 9, 10, 11, 12, 13, 14, 15, and 16). Higher total scores indicate a stronger father-infant bond.

SECONDARY OUTCOMES:
The Behavioral Pediatric Feeding Assessment Scale | 6-month and 9-month infant check-ups
  The Behavioral Pediatric Feeding Assessment Scale (BPFAS), developed by Crist and colleagues and adapted into Turkish by Önal and colleagues, is a 35-item scale. The scale primarily focuses on the child's feeding behavior, with 25 items specifically addressing the child's feeding status. The Turkish adaptation study concentrated solely on these 25 items. Items on the scale are rated on a 5-point Likert scale. Among the 25 items related to children, 6 are positively worded (items 1, 3, 5, 6, 9, and 16) while 19 are negatively worded. Positively worded items are scored in reverse. The minimum possible score on the BPFAS is 35, and the maximum is 175. Higher scores indicate more severe feeding problems and habits. The scale includes four items related to specific feeding difficulties: 'Food selectivity', 'Early food refusal', 'Early refusal of textured foods', and 'Late food refusal'
The Generalized Anxiety Disorder-7 | 6-month and 9-month infant check-ups
  The Generalized Anxiety Disorder-7 Item Scale (GAD-7), developed by Spitzer et al. in 2006 and adapted into Turkish by Konkan et al. in 2011, is a 7-item, 4-point Likert scale designed to assess the severity of generalized anxiety disorder (GAD) over the past two weeks. Cut-off scores of 5, 10, and 15 represent mild, moderate, and severe anxiety, respectively. When a total score cutoff of 10 is used, the scale demonstrates a sensitivity of 89% and a specificity of 82% for diagnosing GAD.
The Edinburgh Postnatal Depression Scale | 6-month and 9-month infant check-ups
  The Edinburgh Postnatal Depression Scale (EPDS), adapted into Turkish by Engindeniz, is a 10-item self-report questionnaire designed to assess symptoms of postnatal depression. Responses are scored on a 4-point Likert scale ranging from 0 to 3, with a total possible score of 30. Items 1, 2, and 4 are scored in a direct manner (0, 1, 2, 3), while items 3, 5, 6, 7, 8, 9, and 10 are reverse-scored (3, 2, 1, 0). A cutoff score of 13 is commonly used to identify women at risk for postnatal depression. Women scoring 13 or above are considered to be at risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Guideline for complementary feeding of infants and young children 6-23 months of age [Internet]. Geneva: World Health Organization; 2023. Available from http://www.ncbi.nlm.nih.gov/books/NBK596427/ PMID 37871145
- [Background] Gökçay G, Keskindemirci G, Mutlu D, Sapmaz S. Basic Information for Families on Child Health and Safety in the First 5 Years. Healthy Nutrition, Istanbul (2021).
- [Background] Onal S, Calık Var E, Uçar A. Adaptation Study of the Behavioral Pediatric Feeding Assessment Scale (BPFAS) into Turkish. Nevşehir Journal of Science and Technology. 2017;6(1):93-101. doi:10.17100/nevbiltek.296685
- [Background] Engindeniz N. Validity and Reliability Study for the Turkish Version of the Edinburgh Postnatal Depression Scale. Unpublished Master's Thesis, Ege University Institute of Health Sciences; 1996.
- [Background] Yilmaz B, Oskay Ü. Karitane Parenting Confidence Scale: Turkish Validity and Reliability Study. Cukurova Medical Journal. 2021;46(2):801-813. doi:10.17826/cumj.902521
- [Background] Güleç D. Examination of the Validity and Reliability of the Father-Infant Attachment Scale in Turkish Society. MS Thesis. Ege University, 2010.
- [Background] Konkan R, Senormanci O, Guclu O, Aydin E, Sungur MZ, Generalized Anxiety Disorder-7 (GAD-7) Test: Turkish Adaptation, Validity and Reliability. Archives of Neuropsychiatry/Noropsychiatri Arsivi 50.1 (2013)
- [Background] Crist W, Dobbelsteyn C, Brousseau AM, Napier-Phillips A. Pediatric assessment scale for severe feeding problems: validity and reliability of a new scale for tube-fed children. Nutr Clin Pract. 2004 Aug;19(4):403-8. doi: 10.1177/0115426504019004403. PMID 16215132
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Crncec R, Barnett B, Matthey S. Development of an instrument to assess perceived self-efficacy in the parents of infants. Res Nurs Health. 2008 Oct;31(5):442-53. doi: 10.1002/nur.20271. PMID 18297638
- [Background] Condon, J. T., Corkindale, C. J., & Boyce, P., (2008). Assessment of postnatal paternal-infant attachment: development of a questionnaire instrument. Journal of Reproductive and Infant Psychology, 26(3), 195-210. https://doi.org/10.1080/02646830701691335
- See also: Konkan R, Senormanci O, Guclu O, Aydin E, Sungur MZ, Generalized Anxiety Disorder-7 (GAD-7) Test: Turkish Adaptation, Validity and Reliability — http://noropsikiyatriarsivi.com/sayilar/415/buyuk/53-58.pdf
- See also: Güleç D. Examination of the Validity and Reliability of the Father-Infant Attachment Scale — http://www.j-humansciences.com/ojs/index.php/ijhs/article/view/2590/1178
- See also: Yilmaz B, Oskay Ü. Karitane Parenting Confidence Scale: Turkish Validity and Reliability Study — http://dergipark.org.tr/tr/pub/cumj/issue/62101/902521
- See also: Onal S, Calık Var E, Uçar A. Adaptation Study of the Behavioral Pediatric Feeding Assessment Scale (BPFAS) into Turkish — http://dergipark.org.tr/en/pub/nevbiltek/issue/28378/296685